CLINICAL TRIAL: NCT07203326
Title: Microsurfaced Acellular Dermal Matrix for Root Coverage Procedures
Brief Title: Microderm for Root Coverage Procedures
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024H0313
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Connective Tissue Graft; Gum Recession
Keywords: Connective Tissue; Wound healing; Tooth root; Mouth; patient comfort; treatment outcome; acellular dermis matrix
MeSH Terms: conditions — Gingival Recession | interventions — Alloderm

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant and blinded evaluator will be not be told which treatment area received which treatment (Alloderm or Microderm). Outcome assessor will not know the group rendering.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- mADM (Experimental): The subjects in this arm will receive microderm as a soft tissue grafting material
  Interventions: Biological: MicroDerm
- ADM (Active Comparator): The patients in this group will receive alloderm as a soft tissue grafting material
  Interventions: Biological: Alloderm

INTERVENTIONS:
Biological: Alloderm — Alloderm is a ready to use tissue graft, made from donated allograft human dermis, processed to remove cells while preserving biologic components and structure of the dermal matrix.
  Other Names: donated allograft human dermis; regenerative tissue matrix
  Arms: ADM
Biological: MicroDerm — MicroDerm is an acellular dermal matrix sourced from donated human tissue. Cytoplast™ MicroDerm is micro-surfaced.
  Other Names: micro-surfaced acellular dermal matrix
  Arms: mADM

SUMMARY:
This randomized pilot study will compare Acellular Dermal Matrix (ADM) and a microsurfaced Acellular Dermal Matrix (mADM) for wound healing, root coverage, gum tissue coverage of the surgical site, blood flow to the site, and patient comfort.

DETAILED DESCRIPTION:
Advancements in Periodontal Surgery techniques and materials have continuously progressed to improve patient dental health. While the patient's own gum tissue from another site of the mouth as a graft [subepithelial connective tissue graft (SCTG)] remains the benchmark for tooth root coverage and increasing gum tissue, there are disadvantages to this surgical method. One disadvantage with this surgical method is the patient will have two surgical sites, one for the graft and one for the coverage of the exposed roots. Another disadvantage, there is limited tissue on the roof of the mouth for covering multiple exposed roots, which means multiple surgeries to cover all the exposed roots. For over 25 years, connective tissue graft surgery using Acellular Dermal Matrix (ADM) has served as an alternative to tissue grafts using the patient's own tissues. ADM is a processed material often used in gum surgery to avoid taking tissue from another part of the mouth) While ADM may not match SCTG for stability and gain in gum tissue, ADM remains a viable alternative to SCTG. Recently, a new ADM [microsurfaced Acellular Dermal Matrix (mADM)] has been developed to enhance healing and improve the surgical outcome. This randomized pilot study will compare ADM and mADM for wound healing, root coverage, gum tissue coverage of the surgical site, blood flow to the site, and patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* Participants 18+ years of age who require a tissue graft due to gum tissue recession.

Exclusion Criteria:

1. Current smokers or users of nicotine replacement products
2. Patients with diabetes (HbA1c > 5.6%)
3. Pregnant or lactating women
4. Surgical sites with previous soft tissue graft.
5. Patients with a history of bisphosphonate therapy, radiotherapy in the head and neck region for malignancies, or chemotherapy for treatment of malignant tumors
6. Patients who are taking anticoagulant and antiplatelet medications.
7. Patients with contraindications, e.g., allergy, for any of the medications used in the study (benzocaine, lidocaine, chlorhexidine rinse, ibuprofen)
8. Poor oral hygiene (PII >2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical root coverage in percentage | From enrollment to up to one year after connective tissue graft surgery.
  To compare the wound healing of root coverage procedures, and the gain of root coverage using either a new microsurfaced Acellular Dermal Matrix(mADM) or Acellular Dermal Matrix (ADM).

SECONDARY OUTCOMES:
Comfort and aesthetic outcome as perceived by patient | From enrollment to up to one year after connective tissue graft surgery.
  By using a Visual Analog Scale (VAS) for Pain and a VAS for aesthetics, patients will note their comfort and appearance of the surgical site at different points after surgery. Scale for pain is from 0 (no pain) to 10 (worse pain imaginable). Scale for aesthetic is 0 (not meeting expectation/unnatural looking/no improvement) to 10 (perfect/natural/significant improvement).

OTHER OUTCOMES:
Blood perfusion in the graft | From enrollment to up to one year after connective tissue graft surgery.
  Through the use of laser speckle contrast imaging (LASCA), the blood perfusion of the surface of the gum tissue/graft area will be recorded. LASCA is a non-invasive technique that maps blood flow in real-time by analyzing the fluctuations in a laser-generated speckle pattern, which is affected by moving red blood cells. This method provides two-dimensional perfusion maps, making it useful for studying and monitoring blood flow in tissues and organs without contrast agents.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University College of Dentistry, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No